CLINICAL TRIAL: NCT02411110
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating Safety and Efficacy of LiRIS® 400 mg in Females With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: A Safety and Efficacy Study of LiRIS® in Females With Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201025-002
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Cystitis, Interstitial; Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2) (Experimental): Treatment Period 1: continuous release of lidocaine inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 1. Treatment Period 2: optional continuous release of lidocaine inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 2.
  Interventions: Combination Product: LiRIS®
- LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2) (Other): Treatment period 1: Matching placebo device to LiRIS inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 1. Treatment Period 2: optional continuous release of lidocaine inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 2.
  Interventions: Combination Product: LiRIS®; Combination Product: LiRIS Placebo

INTERVENTIONS:
Combination Product: LiRIS® — LiRIS® is a drug-device combination product which is placed in the bladder during cystoscopy and remains in the bladder, gradually releasing lidocaine until removed from the bladder via cystoscopy.
Combination Product: LiRIS Placebo — LiRIS placebo is a drug-device combination product, matching the LiRIS® which is placed in the bladder during cystoscopy, remains in the bladder until removed from the bladder via cystoscopy.
  Arms: LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2)

SUMMARY:
This is a safety and efficacy study of LiRIS® in females with interstitial cystitis/bladder pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of interstitial cystitis or bladder pain syndrome

Exclusion Criteria:

* Diagnosis of interstitial cystitis with Hunner's lesions/ulcers
* Previous treatment with LiRIS®

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2017-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Till Geib, Study Director — Allergan
Locations (34):
- United States (31):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - IC Study LLC, Escondido, California
  - Tower Urology, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Genesis Research LLC, San Diego, California
  - Sutter Health, Vacaville, California
  - Women's Health Specialty Care, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - Manatee Medical Research Institute, Bradenton, Florida
  - Atlanta Medical Research Instititute, Alpharetta, Georgia
  - Idaho Urologic Institute, Meridian, Idaho
  - Associated Surgeons and Physicians LLC DBA Women's Health Advantage, Fort Wayne, Indiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Anne Arundel Urology, P.A., Annapolis, Maryland
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Beyer Research, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Washington University, St Louis, Missouri
  - Saint Louis University School of Medicine Department of Obstetrics, Gynecology, and Women's Health Division of Research, St Louis, Missouri
  - Cooper University Hospita/ Univeristy Urogynecology Associates, Voorhees Township, New Jersey
  - Western New York Urology Associates, Cheektowaga, New York
  - BRANY, as agent The Arthur Smith Institute for North Shore Long Island Jewish Health System, Lake Success, New York
  - Urology Institute of Long Island, Plainview, New York
  - McKay Urology, Charlotte, North Carolina
  - Alliance Urology Specialist, P.A., Greensboro, North Carolina
  - Eastern Urological Associates, PA, Greenville, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - MetroHealth System, Cleveland, Ohio
  - Female Sexual and Pelvic Health Institute, Philadelphia, Pennsylvania
  - Integrity Medical Research (Urology Northwest), Mountlake Terrace, Washington
  - University of Washington, Seattle, Washington
- Canada (3):
  - Silverado Research Inc, Victoria, British Columbia
  - Urology Associates/Urologic Medical Research, Kitchener, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario

REFERENCES:
- [Derived] Evans R, Kohan A, Moldwin R, Radecki D, Geib T, Peters KM. Safety, tolerability, and efficacy of LiRIS 400 mg in women with interstitial cystitis/bladder pain syndrome with or without Hunner lesions. Neurourol Urodyn. 2021 Sep;40(7):1730-1739. doi: 10.1002/nau.24702. Epub 2021 Jul 20. PMID 34288094
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, plesase contact IR-CTRegistration@Allergan.com for assistance. — http://www.AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2): Treatment Period 1: LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 1. Treatment Period 2: optional LiRIS® inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 2.
- LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2): Treatment Period 1: Matching placebo device to LiRIS inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 1. Treatment Period 2: optional LiRIS® 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 2.
Period: Treatment Period 1
Arm/Group | LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2) | LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2)
Started | 65 | 66
Completed | 56 | 59
Not Completed | 9 | 7
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Personal Reasons | 2 | 5
Not completed — Other Miscellaneous Reasons | 2 | 0
Period: Treatment Period 2
Arm/Group | LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2) | LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2)
Started | 50 (Period 2 was optional.) | 48 (Period 2 was optional.)
Completed | 49 | 44
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Personal Reasons | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2) | LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2) | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.58 (14.50) | 44.20 (12.65) | 46.37 (13.73)
Age, Customized [Number; unit: participants]
  < 40 Years | 25 | 24 | 49
  ≥ 40 Years | 40 | 42 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 66 | 131
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Average Bladder Pain to Treatment 1 Week 4 Follow-up
Description: The participant recorded their bladder pain over the previous 24-hour period in a 7-day pain assessment tool using an 11-point Numeric Rating Scale (NRS) (0 to 10) where 0=no pain to 10= worst pain. Pain data recorded over the 7-day period were averaged. A negative change from Baseline indicates improvement. An Analysis of Covariance (ANCOVA) model with baseline value as a covariate and treatment group and stratification factors (age group: < 40 years or ≥ 40 years and baseline bladder pain NRS: ≤ 6 or > 6) as factors was used for analysis.
Time Frame: Baseline (Days -7 to 0) to Treatment 1 Week 4
Population: Modified Intent-to-Treat (mITT) Analysis Population included all participants who were randomized and received Treatment 1.
Measure: Least Squares Mean (90% Confidence Interval); unit: score on a scale
Groups:
- LiRIS® (Treatment Period 1): Treatment Period 1: LiRIS® (continuous release of lidocaine ) 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 1.
- LiRIS Placebo (Treatment Period 1): Treatment Period 1: Matching placebo device to LiRIS inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 1.
Arm/Group | LiRIS® (Treatment Period 1) | LiRIS Placebo (Treatment Period 1)
Number analyzed (Participants) | 65 | 66
score on a scale | -1.2 [-1.77 to -0.58] | -1.5 [-2.14 to -0.87]
Statistical Analysis 1: Comparison: LiRIS Placebo (Treatment Period 1); Test type: Superiority or Other; p = 0.505, ANCOVA; Baseline value as a covariate; treatment group and stratification (age: < 40 or ≥ 40 years and baseline bladder pain NRS: ≤ 6 or > 6) as factors; Least Squares Mean Difference = 0.34 — LiRIS® - Placebo

ADVERSE EVENTS:
Groups:
- LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2): Participants who received Matching placebo device to LiRIS inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 1; followed by, LiRIS® (continuous release of lidocaine) 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 2.
- LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2): Participants who received LiRIS® 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 1; followed by, LiRIS® 400 mg inserted into the bladder by cystoscopy on Day 0 and removed on Day 14 of Period 2.
Arm/Group | LiRIS Placebo (Treatment Period 1) | LiRIS® (Treatment Period 1) | LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2) | LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2)
Serious Adverse Events (participants affected / at risk) | 1/66 | 2/65 | 1/48 | 0/50
Other Adverse Events (participants affected / at risk) | 22/66 | 22/65 | 4/48 | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LiRIS Placebo (Treatment Period 1) (N=66) | LiRIS® (Treatment Period 1) (N=65) | LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2) (N=48) | LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2) (N=50)
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pelvic congestion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LiRIS Placebo (Treatment Period 1) (N=66) | LiRIS® (Treatment Period 1) (N=65) | LiRIS Placebo (Treatment Period 1)/LiRIS® (Treatment Period 2) (N=48) | LiRIS® (Treatment Period 1)/LiRIS® (Treatment Period 2) (N=50)
Nausea (Gastrointestinal disorders) | 1 | 4 | 2 | 2
Urinary tract infection (Infections and infestations) | 16 | 10 | 4 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 4 | 3 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 6 | 2 | 0
Dysuria (Renal and urinary disorders) | 11 | 13 | 0 | 2
Urethral pain (Renal and urinary disorders) | 4 | 6 | 3 | 2
Bladder pain (Renal and urinary disorders) | 5 | 4 | 1 | 1
Haematuria (Renal and urinary disorders) | 6 | 2 | 1 | 1
Bladder discomfort (Renal and urinary disorders) | 1 | 5 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 3
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.